CLINICAL TRIAL: NCT01983163
Title: Efficacy of Modified Atkins Diet Versus Ketogenic Diet in Children With Refractory Epilepsy Aged 1 Year to 18 Years: a Randomized Controlled Trial
Brief Title: Dietary Therapy in Children With Refractory Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Addl. Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9968480606
Record Dates: First submitted 2013-11-04; First posted 2013-11-13 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketogenic diet (Active Comparator): ketogenic diet (2.5 to 4:1)
  Interventions: Other: Ketogenic diet (2.5 to 4:1)
- Modifid Atkin's diet (Active Comparator): Modified Atkin's Diet
  Interventions: Other: Modified Atkin's diet

INTERVENTIONS:
Other: Ketogenic diet (2.5 to 4:1) — Minimum ratio (2.5 to4:1) ketogenic diet causing ketosis will be given
  Arms: ketogenic diet
Other: Modified Atkin's diet — 1:1 fixed ketogenic ratio Modified atkins diet will be given
  Arms: Modifid Atkin's diet

SUMMARY:
In children aged 1yr -18 years with refractory epilepsy Modified Atkins diet as add on to ongoing AED therapy would not be inferior compared to ketogenic diet ** in terms of seizure reduction from baseline seizure frequency at 6 months

DETAILED DESCRIPTION:
Primary objective:

To compare the efficacy of Modified Atkins diet compared to Ketogenic diet * in children aged 1 year to 18 years of age with refractory epilepsy on anti epileptic drugs at 6 months of diet intake in terms of percentage of seizure reduction from base line.

Secondary objective:

Proportion of patients who achieve > 50% seizure reduction from baseline after 6 months in both groups To evaluate the nature of adverse events in both the groups

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years with refractory epilepsy*
* Willing to come for regular follow up
* No motivational or psychosocial issues in the family which would preclude compliance with the diet

Exclusion Criteria

* Surgically remediable cause for refractory epilepsy
* Suspected mitochondrial disorder or diagnosed with a disorder in which high fat diet is contraindicated
* Previously received ketogenic diet or modified Atkins diet
* Chronic systemic disease like chronic kidney disease, chronic liver disease, heart disease (congenital and acquired) and chronic respiratory illness

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percentage of seizure reduction at 6 months ( sz frequency / wk average of 4 wks) from base line | Baseline and 6 months
  To develop an optimal dietary therapy for management of refractory epilepsy in children and adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, MD, Principal Investigator — AIIMS, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India